CLINICAL TRIAL: NCT03651882
Title: Intramyometrial and Intravenous Oxytocin Compared to Intravenous Carbetocin for Prevention of Postpartum Hemorrhage in Elective Cesarean Sections - a Monocentric Randomized Controlled Study
Brief Title: Oxytocin i.m./i.v. Versus Carbetocin i.v. in Elective Cesarean Sections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BASEC-Nr: 2017-01750
Record Dates: First submitted 2018-07-24; First posted 2018-08-29 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; carbetocin

STUDY DESIGN:
Intervention Model Description: Before c-section the patients will be randomized to the oxytocin or the carbetocin group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Active Comparator)
  Interventions: Drug: Oxytocin
- Carbetocin (Active Comparator)
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin given in a combined regimen: after delivery 10 IE of oxytocin are applied intramyometrially and 10 IE of oxytocin are given over an infusion of 1000ml of 0.9% NaCL over 12 hours intravenously.
  Arms: Oxytocin
Drug: Carbetocin — Carbetocin is given 0.1mg intravenously as a bolus after delivery.
  Arms: Carbetocin

SUMMARY:
Objective is to proof non-inferiority of intramyometrial and intravenous oxytocin application compared to intravenous carbetocin for prevention of postpartum hemorrhage in planned, uncomplicated cesarean deliveries.

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean section
* present informed consent
* completed 36 weeks of gestation

Exclusion Criteria:

* need for intubation (carbetocin is only licensed for epidural or spinal anesthesia)
* multiple fetus pregnancy
* known coagulopathy
* Placenta praevia
* morbidly adherent placenta
* placental abruption
* thrombocyte dysfunction
* HELLP-syndrome
* preeclampsia
* history of uterine atony

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
incidence of women with a delta hemoglobin ≥ 30g/l. | 48 hours
  Delta hemoglobin is defined as the difference of the hemoglobin at admission minus the hemoglobin after delivery, usually 24-48 hours after the delivery.

SECONDARY OUTCOMES:
adverse maternal outcome parameters | 15 days
  decrease in hemoglobin (delta hemoglobin, in g/l)
adverse maternal outcome parameters | 15 days
  estimated blood loss (in mL),
adverse maternal outcome parameters | 15 days
  incidence of PPH (in %)
adverse maternal outcome parameters | 15 days
  use of additional uterotonic agents (prostaglandines)
adverse maternal outcome parameters | 15 days
  blood transfusion (number of packed red cells)
adverse maternal outcome parameters | 15-300 minutes
  length of surgery (in minutes)
adverse maternal outcome parameters | 15 days
  number of patients with revision (second surgery in the 24hours following the primary cesarean section)
adverse maternal outcome parameters | 15 days
  admission to an intensive care unit (%)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Haslinger, M.D., Study Chair — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided